CLINICAL TRIAL: NCT04166019
Title: Effectiveness of a Peer-led Self-Management Program for People With Recent-onset Psychosis: A Randomized Controlled Trial
Brief Title: Effect of a Peer-led Self-management Program for Recent-onset Psychosis
Acronym: PLSMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Integrated Community Centers for Mental Wellness (Unknown)
Responsible Party: Principal Investigator, Prof. Wai Tong CHIEN, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 19101314
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Early Psychosis; Psychotic Disorders
Keywords: first-onset psychosis; randomized controlled trial; peer support; self management; recovery; re-hospitalization
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment; repeated-measures 3-arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors and researchers (and center staff) are blind to the group assignment and intervention undertaken and concealed to the participant list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Peer-led self-management program (Experimental): Peer-led self-management program (PLSMI) consists of 10 weekly/biweekly, 1.5-hour sessions (4 months), based on the modified Crisis-resolution-team Optimization and Relapse Prevention (CORE) program workbook/manual and psycho-education programs developed by the research team. The program based on completion of a self-management workbook, consisting of the main components: personal recovery goals, plans to re-establish community functioning and support networks following a crisis, identifying early warning signs and creating a relapse prevention plan, and strategies and coping resources to problem-solving and maintain well-being. Participants work through the workbook at their own pace, with the support from the peer support worker, to facilitate/support their recovery. They will meet in group with a trained peer support worker on 10 sessions, usually at 7-12 days intervals over 4 months.
  Interventions: Behavioral: Peer-led self-management program; Behavioral: Usual care
- Psycho-education group (Active Comparator): Psycho-education groups (12-18 members/group; 10 two-hour sessions, weekly/biweekly), 4-month duration similar to the PLSMI, will be led by one trained advanced practice psychiatric nurse in each center experienced in psychiatric rehabilitation, and are guided by a validated group-intervention protocol based on the research team's and McFarlane et al.'s psycho-education programs for psychosis.
  Interventions: Behavioral: Psycho-education group; Behavioral: Usual care
- Usual care only (Other): Usual care (control) participants (and treatment groups) will receive routine psychiatric outpatient and community mental healthcare services.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Peer-led self-management program — The program based on completion of a self-management workbook, consisting of the main components: personal recovery goals, plans to re-establish community functioning and support networks following a crisis, identifying early warning signs and creating a relapse prevention plan, and strategies and coping resources to problem-solving and maintain well-being.
  Other Names: PLSMI
  Arms: Peer-led self-management program
Behavioral: Psycho-education group — The psycho-education group program is comprised of six components: introduction and goal-setting; basic understanding of psychosis and symptom and emotion self-care; education workshop of psychosis care, treatment and community support services; learning about self-care skills; establishing social support and effective coping skills; and skills practices, review and future plan.
  Arms: Psycho-education group
Behavioral: Usual care — Routine care services consist of monthly psychiatric consultation and treatments prescribed by psychiatrist, nursing advice on community care, brief education (1-2 hourly sessions) about mental illness/treatments by psychiatric nurses, home visits by case managers, and/or referrals to community/welfare services.

SUMMARY:
This randomized controlled trial is to test the effectiveness of a peer-led self-management program (PLSMI) for people with recent-onset psychosis in the community over 18-month follow-up, compared with a conventional psychoeducation group and routine community mental healthcare.

DETAILED DESCRIPTION:
Objectives: to investigate the effectiveness of a peer-led self-management intervention (PLSMI) for recent-onset psychosis on patient outcomes over 18-months follow-up, compared with a conventional psycho-education group and routine care only group.

Hypotheses: When compared with those in a psycho-education group and routine care, the PLSMI participants will indicate significantly greater:

1. Improvement in patients' level of recovery at 1-2 weeks post-intervention (Primary hypothesis and outcome);
2. Reduction of their re-hospitalization rates and symptom severity, and/or improvement in functioning, satisfaction with service, problem-solving, and insight into illness at 1-2 weeks post-intervention; and/or
3. Improvements in the above outcomes (hypotheses 1) at 6-, 12- and/or 18-month follow-ups.

Primary outcome is patients' level of recovery. Qualitative interviews with purposely selected PLSMI participants and all peer support workers (agreed for interview) will enhance understanding about their perceived benefits, service satisfaction, strengths, and limitations of the intervention undertaken from peer-workers' and participants' perspectives.

Study Design: A multi-center randomized controlled trial with repeated-measures, three-group design on a community-based PLSMI will be conducted with both outcome and process evaluation.

Subjects: 180 people with recent-onset psychosis (not more than 3 years onset) randomly selected from 6 Integrated Community Centers for Mental Wellness and randomly assigned into 3 arms.

Instruments/Measures: Level of self-reported recovery (QPS, primary outcome); occurrence and frequency of and time to psychiatric hospitalization over past 6 or 18 months; symptom severity (PANSS); problem solving ability (C-SPSI-R:S); illness insight (ITAQ); functioning (SLOF), and service satisfaction (CSQ-8).

Focus group interviews will be conducted to collect views on benefits and weaknesses of PLSMI.

Data analyses: Comparing the mean value changes of outcomes between-groups across time on intention-to-treat basis, using MANOVA/Mixed Modeling/Generalized Estimation Equations test and comparing the occurrence of and time to hospitalization between groups using survival analysis and Cox regression test; content analysis of qualitative data from focus-group interviews and intervention sessions.

Expected results: The findings provide evidence of the effectiveness of peer-support self-management program for early-stage psychosis in community mental health healthcare on improving patients' recovery and other important patient outcomes, as well as service satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese residents, aged 18-60 years;
* Having Global Assessment of Functioning scores ≥ 51, indicating mild to moderate symptoms and difficulty in psychosocial/occupational functioning and thus mentally stable to comprehend the self-care training and education provided; and
* Able to understand Cantonese/Mandarin

Exclusion Criteria:

* Participated in or having been receiving other psycho-education/psychotherapies;
* Having co-morbidity of another mental illness (learning disability and cognitive and personality disorders) or any clinically significant medical diseases; and
* Having visual/language/communication difficulty

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire about the Process of Recovery (QPR) | At recruitment
  Level of recovery from illness is measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). Items are rated on a 5-point Likert scale (0=disagree strongly to 4=agree strongly; score range= 0-88); the higher total score indicates a higher of recovery progress.
Questionnaire about the Process of Recovery (QPR) | At 1-2 weeks post-intervention
  Level of recovery from illness is measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). Items are rated on a 5-point Likert scale (0=disagree strongly to 4=agree strongly); the higher total score indicates a higher of recovery progress.
Questionnaire about the Process of Recovery (QPR) | At 6 months post-intervention
  Level of recovery from illness is measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). Items are rated on a 5-point Likert scale (0=disagree strongly to 4=agree strongly); the higher total score indicates a higher of recovery progress.
Questionnaire about the Process of Recovery (QPR) | At 12 months post-intervention
  Level of recovery from illness is measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). Items are rated on a 5-point Likert scale (0=disagree strongly to 4=agree strongly); the higher total score indicates a higher of recovery progress.
Questionnaire about the Process of Recovery (QPR) | At 18 months post-intervention
  Level of recovery from illness is measured with the Questionnaire about the Process of Recovery (QPR) developed by Neil et al. (2009). Items are rated on a 5-point Likert scale (0=disagree strongly to 4=agree strongly); the higher total score indicates a higher of recovery progress.

SECONDARY OUTCOMES:
Re-hospitalization rate | Change from recruitment to 18 months follow-up
  Occurrence of and time to hospitalization, and frequency of re-hospitalizations over past 5-6 months
Positive and Negative Syndrome Scale (PANSS) | Change from recruitment to 18 months follow-up
  Symptom severity is assessed with the 30-item Positive and Negative Syndrome Scale (PANSS) developed by Kay (1987) across three sub-scales: positive symptoms, negative symptoms and general psychopathology. Items are rated on a 7-point Likert scale (1= absent to 7= extreme; total score range= 7-210); a higher total score indicates more severe psychotic symptoms.
Specific Level of Functioning Scale (SLOF) | Change from recruitment to 18 months follow-up
  Patient functioning is measured by the 43-item Specific Level of Functioning Scale (SLOF) developed by Schneider and Struening (1983) in terms of three domains: physical functioning/personal care, social functioning and community living skills. Items are rated on a 5-point Likert scale (1=very poor to 5=very well; total score range= 43-215); a higher total score indicates a higher level of functioning.
Revised Social-Problem-Solving Inventory (C-SPSI-R:S) | Change from recruitment to 18 months follow-up
  Problem-solving ability will be assessed with a 25-item Chinese version of Revised Social-Problem-Solving Inventory (C-SPSI-R:S), comprising 2 domains: problem-solving style (rational/impulsive; careless/avoidance) and orientation (positive/negative). Items are rated on a 5-point Likert scale (1=not at all true to 4=extremely true; total score range= 0-100); a higher total score indicates better problem solving ability.
Insight and Treatment Attitude Questionnaire (ITAQ) | Change from recruitment to 18 months follow-up
  Insight into illness and treatment is measured by the 11-item Treatment Attitude Questionnaire (ITAQ) developed by McEvoy et al. (1989) measuring patients' insights and recognition of their illness and attitudes towards the need for treatments. Items are rated on a 3-point Likert scale (0=not necessary to receive treatment to 2=treatment should be required/continued regularly; total score range= 0-22; a higher total score indicates better insight into the illness/treatment.
Client Satisfaction Questionnaire (CSQ-8) | Change from recruitment to 18 months follow-up
  Patient satisfaction with service is measured by the 8-item Client Satisfaction Questionnaire (CSQ-8) developed by Attkisson and Zwick (1982). Items are rated on a 4-point Likert scale (1= very dissatisfied to 4= very satisfied; total score range= 8-32); a higher total score indicates a better satisfaction with the services received/receiving.

CONTACTS AND LOCATIONS:
Overall Officials: Wai Tong Chien, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Integrated Community Centers for Mental Wellness, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The name and email of the researchers can be shared openly for communication and collaboration.

REFERENCES:
- [Background] Johnson S, Lamb D, Marston L, Osborn D, Mason O, Henderson C, Ambler G, Milton A, Davidson M, Christoforou M, Sullivan S, Hunter R, Hindle D, Paterson B, Leverton M, Piotrowski J, Forsyth R, Mosse L, Goater N, Kelly K, Lean M, Pilling S, Morant N, Lloyd-Evans B. Peer-supported self-management for people discharged from a mental health crisis team: a randomised controlled trial. Lancet. 2018 Aug 4;392(10145):409-418. doi: 10.1016/S0140-6736(18)31470-3. PMID 30102174
- [Background] Chien WT, Bressington D, Chan S, Lubman DI. Effects of peer-support illness-management program for people with recent-onset psychosis (Oral presentation, Proceeding p. 14). THE IRES - 627TH INTERNATIONAL CONFERENCES ON ECONOMICS AND SOCIAL SCIENCES (ICESS; June 2019). Thailand: Bangkok.